CLINICAL TRIAL: NCT04636320
Title: Prevalence of Silent Myocardial Scars on Cardiac Magnetic Resonance Following COVID-19 Infection
Brief Title: Prevalence of Myocardial Scars on CMR After COVID-19 Infection
Acronym: COVID-CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Grant Agreement ERC n°715093 (Unknown); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2020/22
Record Dates: First submitted 2020-11-18; First posted 2020-11-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Virus Disease
Keywords: Myocardial Scar; Cardiac Magnetic Resonance; Arrhythmia
MeSH Terms: conditions — COVID-19; Virus Diseases; Arrhythmias, Cardiac | interventions — Blood Specimen Collection; Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: Single-centre case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group COVID-19 (Experimental): 120 patients with history of laboratory-proven symptomatic COVID-19 infection managed without hospitalization
  Interventions: Device: Contrast-enhanced CMR; Diagnostic Test: Exercise test ECG; Biological: Blood sample; Diagnostic Test: Resting 12 lead ECG; Diagnostic Test: 24 hour Holter ECG
- Healthy volunteer group (Active Comparator): 120 healthy volunteers. Age- and sex-matched controls
  Interventions: Device: Contrast-enhanced CMR; Diagnostic Test: Exercise test ECG; Biological: Blood sample; Diagnostic Test: Resting 12 lead ECG; Diagnostic Test: 24 hour Holter ECG

INTERVENTIONS:
Device: Contrast-enhanced CMR — Cardiac Magnetic Resonance Imaging (MRI) examinations will be performed at Day 0 visit on clinical systems 1.5 equipped with specific antennas for cardiac imaging. The imaging protocol will last approximately 50 minutes.
Diagnostic Test: Exercise test ECG — A treadmill exercise test with 12 lead ECG monitoring will be performed at M3 visit.
  Maximum expected enrollment 30 MRI+ patients and 30 healthy volunteers MRI- matched controls.
Biological: Blood sample — A blood sample will be taken at Day 0 visit for COVID-19 serology, hematocrit measurement, ultra-high sensitive troponin test, low grade markers of inflammation, genetic profiling.
  An other blood sample will be taken at M3 visit for a control COVID-19 serology for 30 healthy volunteers.
Diagnostic Test: Resting 12 lead ECG — A resting 12 lead ECG will be performed at Day 0 visit.
Diagnostic Test: 24 hour Holter ECG — A 24 hour Holter ECG will be performed at M3 visit. Maximum expected enrollment 30 MRI+ patients and 30 healthy volunteers MRI- matched controls.

SUMMARY:
The aim of this study is to assess the prevalence and arrhythmogenic role of occult myocardial scars on Cardiac Magnetic Resonance (CMR) in a population of patients with history of laboratory-proven symptomatic COVID-19 infection managed without hospitalization, as compared to a population of age- and sex-matched healthy volunteers.

DETAILED DESCRIPTION:
Multiple large series conducted in hospitalized patients have reported high rates of myocardial injuries in the acute stage of COVID-19 infection. These findings have raised concerns regarding potential long term consequences of the pandemic on cardiovascular diseases (heart failure and sudden cardiac deaths due to scar-related arrhythmias). However, the prevalence of silent myocardial injuries in the general population who presented a COVID-19 infection managed without hospitalization are unknown. In addition, the propensity of these scars to generate arrhythmias have not been thoroughly studied. COVID CMR will include 120 patients with history of laboratory-proven symptomatic COVID-19 infection managed without hospitalization and 120 age- and sex-matched controls. At day 1, all subjects will undergo a 12-lead electrocardiogram, a contrast-enhanced CMR study including advanced methods to detect silent myocardial scars, and a blood sample to look for markers of inflammation and cardiac injury, and to assess the COVID-19 serological status at the time of the CMR study. The prevalence of myocardial scars on CMR will be compared between the 2 groups. In a second visit at 3 months, patients showing myocardial scar on CMR will be matched to healthy volunteers showing no such scars, and these 2 population subsets will undergo exercise electrocardiogram (ECG) and 24 hour Holter ECG to characterize the arrhythmogenic role of silent myocardial scars.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 18 years old
* Affiliated to a health insurance program
* Providing free, informed, written and signed consent to participate (at the latest on the day of inclusion and before any research procedure is initiated)
* Effective contraception if women in the age to procreate
* In the patient group : history of COVID-19 infection with either a positive Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) test on nasopharyngeal swab or a positive COVID-19 serology in the acute stage. Presence of all following symptoms in the acute stage: fever>38°C, asthenia, arthromyalgia, associated with at least 2 of the following: coughing and/or spitting, dyspnea and/or chest discomfort, anosmia and/or ageusia.

Exclusion Criteria:

* age < 18 years old
* History of cardiac disease or acute coronary syndrome associated with troponin rise
* History of allergic reaction to gadolinium-based contrast agents
* History of severe renal failure
* Presence of a pacemaker, implantable defibrillator, intra-orbital metallic material, intra-cranial surgical clip, valve prosthesis Star-Edwards pre 6000, neurostimulator or implantable insulin pump
* Claustrophobia or inability to lay on the back for 50 min
* Pregnant or breast feeding women
* Inability to express informed consent
* Person deprived of liberty by judicial or administrative decision
* Person under legal protection
* In the healthy volunteer group:

  * Symptoms suggestive of COVID-19 infection over the epidemic period (after February 1st 2020)
  * Person not willing to be informed of potential incidental CMR findings
* In the patient group:

  * Hospitalization for infectious syndrome suggestive of COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of myocardial scars | Day 0
  Expressed in percentage of participant, as assessed on late gadolinium-enhanced magnetic resonance acquired at high resolution using a free breathing 3D method.

SECONDARY OUTCOMES:
CMR feature : Location and size of myocardial scars | Day 0
  Measured in mL
CMR feature : native T1 and T2 values | Day 0
  Measured in milliseconds
CMR feature : extracellular volume fraction | Day 0
  Measured in percentage
CMR feature : ventricular volumes | Day 0
  Measured in mL/m2
CMR feature : ejection fraction | Day 0
  Measured in percentage
CMR feature : myocardial strain | Day 0
  Measured in percentage
ECG features | Baseline and month 3
  Repolarization abnormalities, T wave inversion, ST segment abnormalities, QRS fractionation, atrial arrhythmias, premature ventricular beats or ventricular tachycardia.These will be assessed at the time of CMR study on a resting 12-lead ECG recording and on exercise 12-lead ECG and 24-hour Holter ECG recordings.
Biological feature : positivity of COVID-19 serology | Baseline and month 3
  Rate of seropositivity in asymptomatic volunteers and rate of seronegativity in patients with a history of symptomatic episodes.
  Measured in percentage.
Biological feature : troponin level | Day 0
  Measured in fg/ml
Biological feature : inflammatory markers level | Day 0
  Markers of inflammation and fibrosis will be sought. The Th1/Th2/activation/inflammation/apoptosis markers will be measured in the sera by a Luminex test allowing the detection of 48 analytes.
Genetic profile research | Day 0
  Identified by sequencing genetic variants that could have an impact on the occurrence of a severe form in individuals infected with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Hubert COCHET, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France